CLINICAL TRIAL: NCT03381755
Title: Comparative Effectiveness and Safety Analysis of Low-dose and Standard-dose Ticagrelor in Chinese Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention
Brief Title: Low-dose Ticagrelor in Chinese ACS Patients Undergoing PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACS-3
Record Dates: First submitted 2017-12-14; First posted 2017-12-22 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2017-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- half-dose ticagrelor (Experimental)
  Interventions: Drug: half-dose ticagrelor
- standard-dose ticagrelor (Active Comparator)
  Interventions: Drug: standard-dose ticagrelor

INTERVENTIONS:
Drug: half-dose ticagrelor — To observe the effectiveness and safety of ticagrelor 45mg bidpo. in Chinese ACS patients undergoing PCI.
  Arms: half-dose ticagrelor
Drug: standard-dose ticagrelor — To observe the effectiveness and safety of ticagrelor 90mg bidpo. in Chinese ACS patients undergoing PCI.
  Arms: standard-dose ticagrelor

SUMMARY:
Dual Antiplatelet Therapy (DAPT) with aspirin and P2Y12 receptor inhibitor remains a cornerstone in the secondary prevention of coronary artery disease (CAD). Clopidogrel is one of the most commonly used antithrombotic agent that inhibits the platelet P2Y(12) adenosine diphosphate (ADP) receptor.

Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for ACS patients. The previous studies have reported that half-dose ticagrelor had the similar inhibitory effect on platelet aggregation as the standard-dose ticagrelor, which was significantly stronger than that in the clopidogrel group. One-quarter standard-dose ticagrelor provided greater degree of platelet inhibition than standard dose clopidogrel in Chinese patients with stable CAD. But the effectiveness and safety of low-dose ticagrelor remain yet not very clearly in Chinese patients with acute coronary syndrome undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* After half-dose ticagrelor (loading dose 90mg, and then 45mg bidpo.) treatment for 3 days, the platelet aggregation is effectively inhibited by light transmission aggregometry method and thromboela-stogram.
* planned to undergo PCI recently
* planned to DAPT for 1 year after PCI

Exclusion Criteria:

* taken adenosine diphosphate (ADP) receptor antagonists within 2 weeks
* Platelet count <100g/L;
* A history of bleeding tendency;
* Aspirin, ticagrelor or clopidogrel allergies;
* Severe liver injury.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-14 (Estimated); Study Completion 2020-12-14 (Estimated)

PRIMARY OUTCOMES:
thromboela-stogram | up to 6 months
  inhibition of platelet aggregation (ADP) ; MA (ADP)
thromboela-stogram | up to 1 year
  inhibition of platelet aggregation; MA

SECONDARY OUTCOMES:
MACE | up to 1 year
  cardiovascular death, non-fatal myocardial infarction and stroke
Side effects including bleeding and dyspnea | up to 1 year
The rate of treatment interruption due to ticagrelor intolerance. | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, PhD, Principal Investigator — Cardiovascular Department, the First Affiliated Hospital of Harbin Medical University
Locations (1):
- Thromboela-Stogram, Beijing, Beijing Municipality, China